CLINICAL TRIAL: NCT06646068
Title: Refining Clinical Judgment Competence in Nursing Education: The Impact of the Philips 66 Brainstorming Technique in Case-Based Learning
Brief Title: Enhancing Clinical Judgment Competence in Nursing Education: A Mixed-Methods Study in the Philippines
Acronym: MMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angeles University Foundation (Other)
Responsible Party: Principal Investigator, Rudena A. Madayag, Assistant Professor, Angeles University Foundation
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-CON-Faculty-002; 2024-CON-Faculty-002 (Other: Angeles University Foundation Ethics Review Committee)
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Clinical Competence; Nursing Education
Keywords: Clinical Judgment Competence in Nursing

STUDY DESIGN:
Intervention Model Description: The study evaluated the effectiveness of the Philips 66 brainstorming technique integrated with case-based learning to enhance clinical judgment competence in nursing students. Using a true experimental pre-test/post-test design, 60 students were randomly assigned to intervention and control groups. Both groups were exposed to the same clinical case scenarios, but the intervention group participated in Philips 66 sessions. The process included individual reflection (6 minutes) on clinical judgment and disaster triage protocols, followed by 6-minute group brainstorming sessions to collaboratively refine ideas. Group leaders then presented their nursing care plans within a 6-minute timeframe. The model aimed to foster critical thinking, collaboration, and clinical decision-making skills. The Lasater Clinical Judgment Rubric (LCJR) was used for evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Philips 66 Brainstorming Technique Group (Intervention Group) (Other): Participants in this group will engage in the Philips 66 Brainstorming Technique as part of their case-based learning sessions. This structured method involves dividing participants into smaller groups of 6, with each group discussing a topic for 6 minutes, aimed at enhancing critical thinking and clinical judgment skills in nursing students.
  Interventions: Other: Philips 66 with CBL

INTERVENTIONS:
Other: Philips 66 with CBL — Each team is given six minutes to brainstorm ideas or solutions to specific clinical cases. This technique is applied during case-based learning sessions to enhance clinical judgment and critical thinking skills among nursing students.
  Other Names: Brainstorming Technique

SUMMARY:
The goal of this mixed-methods study is to assess the impact of the Philips 66 brainstorming technique integrated with case-based learning (CBL) on refining clinical judgment competence in senior nursing students in the Philippines.

The main question it aims to answer is:

Does the Philips 66 technique improve clinical judgment competence among nursing students more effectively than traditional CBL methods?

Participants will be senior nursing students, randomly assigned to an intervention group using the Philips 66-CBL and a control group using standard CBL. Clinical judgment competence will be evaluated through pre- and post-test assessments using the Lasater Clinical Judgment Rubric (LCJR) and confidence questionnaires. A subset of participants from the intervention group will take part in focus group discussions to explore their experiences with the Philips 66 technique. Data will be collected over a short-term period for quantitative and qualitative analysis.

DETAILED DESCRIPTION:
This study utilizes an explanatory sequential mixed-methods design to evaluate the effectiveness of the Philips 66 brainstorming technique, integrated with case-based learning (CBL), in enhancing clinical judgment competence among senior nursing students in the Philippines. The study consists of two phases: a quantitative experimental phase and a qualitative exploratory phase.

The quantitative phase adopts a true experimental pre-test/post-test design, involving 60 senior nursing students who will be randomly assigned to either the intervention group (n=30) or the control group (n=30). The intervention group will undergo CBL sessions facilitated by the Philips 66 technique, while the control group will follow the standard CBL approach. The Philips 66 technique is a structured form of small group brainstorming where participants collaborate in smaller teams, fostering idea generation and peer learning in a timed setting. Clinical judgment competence will be assessed before and after the intervention using the Lasater Clinical Judgment Rubric (LCJR), which measures four dimensions of clinical judgment: noticing, interpreting, responding, and reflecting. Additionally, a researcher-designed questionnaire will be used to measure students' confidence levels in their clinical decision-making abilities.

The qualitative phase will involve focus group discussions (FGDs) with a subset of participants from the intervention group to gain deeper insights into their experiences with the Philips 66 technique. These discussions will aim to explore how the technique influences their critical thinking, decision-making, and collaborative learning processes. Thematic analysis will be applied to identify recurring themes and key experiences.

Statistical analysis for the quantitative component will include descriptive statistics, non-parametric tests (such as the Mann-Whitney U test), and Wilcoxon signed-rank tests to analyze differences in clinical judgment competence and confidence levels between the two groups. For the qualitative component, data from FGDs will be analyzed thematically to provide contextual understanding and support for the quantitative findings.

The study aims to determine whether the integration of the Philips 66 technique with CBL can significantly enhance the development of clinical judgment competence in nursing students, preparing them for the challenges of real-world clinical settings. Future studies may be conducted across different contexts to validate the long-term effects of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* BSN students enrolled in their fourth year at a Higher Education Institution in Angeles City, Philippines.
* At least 20 years old.
* Willing to participate in both pre- and post-intervention assessments.

Exclusion Criteria:

* Undergraduate nursing students who do not meet the criteria and refuse to join the study
* Students with anticipated absences exceeding a certain threshold (e.g., more than two sessions)

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Judgment Competence | Assessment of clinical judgment competence will occur at baseline (pre-intervention) and immediately after the intervention using the Lasater Clinical Judgment Rubric (LCJR) over a one-month period.
  The measure will assess the change in clinical judgment competence using the Lasater Clinical Judgment Rubric (LCJR) pre-intervention and immediately post-intervention.

SECONDARY OUTCOMES:
Change in Teamwork and Collaborative Learning | Focus group interviews to assess teamwork and collaborative learning will be conducted immediately following the intervention, with each interview expected to last approximately 30-60 minutes.
  This measure will evaluate the change in teamwork and collaborative learning as assessed through focus group interviews conducted immediately after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rudena A Madayag, MAN, Principal Investigator — Angeles University Foundation
Locations (1):
- Angeles University Foundation, Mac Arthur Highway, Angeles City, Pampanga, Philippines

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data (IPD) will be shared in this study:
  De-identified Clinical Judgment Competence Scores:
  Pre-test and post-test scores measured using the Lasater Clinical Judgment Rubric (LCJR).
  These scores will be anonymized to protect participants' identities.
  Demographic Data:
  Age, gender, academic year, and other relevant participant characteristics, provided they do not compromise anonymity.
Supporting Information: SAP
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Access Criteria for Sharing IPD and Supporting Information:
  With Whom: IPD and supporting information will be shared with researchers, academic institutions, and healthcare professionals who are engaged in scientific, clinical, or educational research relevant to nursing education and clinical judgment competence. Requests from individuals or organizations with a valid research purpose will be considered.
  Types of Analyses: The shared data can be used for secondary analyses, including but not limited to meta-analyses, replication studies, and the exploration of interventions to improve clinical judgment and reasoning in nursing students. The data can also be used for educational purposes in developing innovative teaching strategies or curricula.
  Mechanism of Access: Requests for access to the data must be submitted in writing to the study's principal investigator. The requests should detail the intended use of the data, the scope of the analyses, and any related publication plans.

REFERENCES:
- [Derived] Madayag RA, Bautista EC, Pineda JPC, Geanga AS, Agustin RMS, Roque ML, Apostol AP, Ramirez DQ. Refining clinical judgment competence in nursing education in the Philippines: A mixed-methods study on the impact of the Philips 66 brainstorming technique in case-based learning. Belitung Nurs J. 2024 Nov 24;10(6):680-694. doi: 10.33546/bnj.3560. eCollection 2024. PMID 39601025